CLINICAL TRIAL: NCT05887180
Title: PräVaNet - Structured, Intersectoral, Multiprofessional, Digitized Program to Optimize Cardiovascular Prevention
Acronym: PräVaNet
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Association of Statutory Health Insurance Physicians (KV Berlin) (Unknown); Statutory health insurance provider AOK Nordost (Unknown); German Foundation for the Chronically ill (DScK) (Unknown); aQua - Institute for Applied Quality Improvement and Research in Health Care GmbH (Unknown); Scientific Institute for Health Economics and Health System Research (WIG2) (Unknown)
Responsible Party: Principal Investigator, Dr. med. David Sinning, Dr. med., German Heart Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 01NVF20001
Record Dates: First submitted 2023-04-05; First posted 2023-06-02 (Actual); Last update posted 2023-06-07 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes; Arteriosclerosis; Arterial Hypertension; Lipid Metabolism Disorders
Keywords: E-Health; Telemedicine; Prevention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Arteriosclerosis; Hypertension; Lipid Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned to 1 of 2 possible treatment arms (standard of care vs. intervention)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PräVaNet-Intervention (Experimental): Interdisciplinary Online-Board, close patient care by a specially trained nurse, E-Health-platform with physician cockpit, patient App, sensor kit (ECG-capable pulse watch, digital blood pressure monitor, digital blood glucose meter if required) and a telemonitoring/alarm system.
  Interventions: Other: PräVaNet-Intervention
- Standard of Care (No Intervention): Standard of Care according to currently valid guidelines.

INTERVENTIONS:
Other: PräVaNet-Intervention — interdisciplinary and digitally supported prevention concept
  Arms: PräVaNet-Intervention

SUMMARY:
PräVaNet is a prospective, 1:1 randomized, controlled trial to investigate the efficacy of a new, digitalized prevention strategy ("ePrevention") in cardiovascular high-risk patients with type 2 diabetes mellitus in the outpatient sector.

DETAILED DESCRIPTION:
PräVaNet is an interdisciplinary and digitally supported prevention concept based on a specialist online board, close patient care by a specially trained nurse, an E-Health platform with physician cockpit, patient App, a smart sensor kit (ECG-capable pulse watch, digital blood pressure monitor, digital blood glucose meter if required) and a telemonitoring/alarm system.

The aim of PräVaNet is to prevent a worsening of the condition of cardiovascular high-risk patients with type 2 diabetes through intensified and continuous risk factor monitoring as well as guideline- and needs-based patient treatment and care. Serious, cost-intensive (especially cardiovascular) secondary diseases are to be avoided and the quality of life of those affected is to be maintained or improved. PräVaNet includes intensive patient education to improve personal responsibility and self-management of the disease and the individual cardiovascular risk.

PräVaNet is the first clinical study evaluating effectiveness and safety of an ePrevention-concept in cardiovascular high-risk patients with type 2 diabetes mellitus in Germany.

ELIGIBILITY:
Inclusion Criteria:

Included are patients who at baseline:

* Are at least 18 years or older
* Living in the German federal states of Berlin or Brandenburg
* Insured by the cooperating German SHI company
* Diagnosed with type 2 diabetes mellitus at least 3 months prior to study entry and who
* Require drug therapy for diabetes mellitus type 2; i.e., received at least 1 oral antidiabetic drug or insulin therapy for at least 3 months prior to study entry; such a need for drug therapy should also exist at the start of the study for the next year and beyond

and

* Fulfill at least one of the following criteria:

  1. metabolic syndrome: 3 of the following 4 criteria: Waist-to-hip ratio (WHR) > 94 cm/80 cm; triglycerides ≥ 150 md/dl or cholesterol- or lipid-lowering therapy; high density lipoprotein (HDL) < 40/50 mg/dl or cholesterol- or lipid-lowering therapy; hypertension ≥ 135/85 mmHg or antihypertensive therapy;

     and/or
  2. macrovascular manifestations (coronary artery disease (CAD) and/or peripheral arterial disease (CAD) and/or carotid stenosis)

     and/or
  3. microvascular manifestation (chronic renal failure with estimated glomerular filtration rate (eGFR) < 60ml/min/1.73m2).

     Exclusion Criteria:

     Patients with at least one of the following characteristics are excluded from participation:
* Chronic disease and, in this context, an anticipated life expectancy of less than 21 months;
* Renal failure requiring dialysis;
* Lipid metabolism disorder and indication for lipid apheresis;
* Mental illness requiring therapy;
* Lack of ability to use E-Health technologies;
* Participation in another intervention study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 209 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adverse cardiovascular and cerebrovascular events (MACCE "Plus" events) | 20 months
  MACCE "Plus" is defined as an index derived from the incidence of major cardiovascular complications (acute coronary syndrome, stroke/transient ischemic attack), death of any etiology, and unplanned hospitalization for any of the following discharge diagnoses: Hyper-glycemia, Hypoglycemia, Amputation, Ischemic Gangrene, Acute Renal Failure with/without Dialysis Requirement, Heart Failure Decompensation, Coronary Revascularization for Unstable Angina.

SECONDARY OUTCOMES:
Cardiovascular risk | 20 months
  A change in the prevalence and treatment quality of cardiovascular risk factors according to a change in the Framingham Risk Score and according to the prevalence of the individual risk factors.
Complication rate | 20 months
  e.g., atrial fibrillation, hypoglycemia, diabetic nephropathy
Adherence to therapy | 20 months
  assessment of medication adherence and assessment of adherence with dietary and exercise measured on a scale from 1=not adherent to 10=fully adherent
Changes in self-reported quality of life | 20 months
  Changes in self-reported quality of life, assessed by the EQ-5D-5L. The EQ-5D-5L consists of 5 dimensions (mobility, self-care, usual activities, pain or discomfort, and anxiety to depression measured on a five-point scale describing the degree of problems in that area (1-no problems to 5-very severe problems)) and results in a single index.
Changes in patient reported quality of care | 20 months
  Changes in patient reported quality of care, measured by the Patient Assessment of Chronic Illness Care (PACIC-5A): 26 items questionnaire measured on a likert scale ranging from min: 1 to max: 5, assessing the patient's perception of greater involvement and receipt of chronic care counseling according to the Chronic Care Model. Higher scores indicate higher quality of care.
Changes in patient reported physical, psychological and social health | 20 months
  Changes in patient reported physical, psychological and social health by using the Patient-Reported Outcomes Measurement Information System (PROMIS®): pain intensity (0-10 numeric rating item) and seven health domains (physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain, each measured on a likert scale of answers ranging from 1-5. The values of all item responses are averaged to generate subscores for each dimension. From these subscores, a global physical health score and a global mental health score are generated. The scores are translated into T-scores according to a reference population with a mean of 50 and a standard deviation of 10. The higher the T-score points, the better the health status.
Changes in diabetes self-care activities | 20 months
  Changes in diabetes self-care activities, measured by the Diabetes Self-Management Questionnaire (DSMQ): scale min = 1; scale max = 4; higher scores mean better treatment behavior
Inpatient health care utilization | 20 months
  Measured by % of patients with hospitalizations/utilized inpatient health care services assessed by SHI data.
Direct medical costs of intervention and control group patients | 20 months
Relative share of outpatient costs, inpatient costs and pharmaceutical costs in total direct medical costs | 20 months
Costs of work incapacity / early retirement of intervention and control group patients | 20 months
Incremental cost-effectiveness ratio (ICER) using the primary outcome measure (MACCE "Plus" events) as the effectiveness criterion (cost-effectiveness analysis) | 20 months
Incremental cost-utility relation (societal perspective) | 20 months
  cost-utility analysis: incremental cost-utility ratio using health-related quality of life as utility (complemented by length of health state for calculation of quality-adjusted-life-years (QALYs))

CONTACTS AND LOCATIONS:
Overall Officials: David Sinning, MD, Principal Investigator — Deutsches Herzzentrum der Charité; Department of Cardiology, Angiology and Intensive Care Medicine
Locations (1):
- Deutsches Herzzentrum der Charité; Department of Cardiology, Angiology and Intensive Care Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Project website — https://kardio-cbf.charite.de/forschung/innovationsfonds_projekt_praevanet/